CLINICAL TRIAL: NCT04765059
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Platinum Plus Pemetrexed Chemotherapy Plus Osimertinib Versus Platinum Plus Pemetrexed Chemotherapy Plus Placebo in Patients With EGFRm, Locally Advanced or Metastatic NSCLC Who Have Progressed Extracranially Following First-Line Osimertinib Therapy (COMPEL)
Brief Title: A Study to Evaluate Chemotherapy Plus Osimertinib Against Chemotherapy Plus Placebo in Patients With Non-small Cell Lung Cancer (NSCLC)
Acronym: COMPEL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5162C00042; 2019-003969-18 (EudraCT Number)
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Osimertinib; Platinum; Pemetrexed; Epidermal growth factor receptor mutation positive (EGFRm); Extracranial progression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, the Investigator, the study team (Sponsor, Contract research organization) and the study site staff will be blinded to osimertinib or placebo allocation. Patients may participate in the open label part of trial at the discretion of the investigator to receive osimertinib and continue any ongoing chemotherapy if intracranial progression is their first progression event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental): All randomized patients will receive osimertinib 80 mg QD with pemetrexed (500 mg/m^2) (with pre-treatment) plus either cisplatin (75 mg/m^2) or carboplatin ([AUC] 5), both administered on Day 1 of 21-day cycles for 4 cycles, followed by osimertinib 80 mg QD plus pemetrexed maintenance (500 mg/m^2) on Day 1 of 21-day cycles
  Interventions: Drug: Osimertinib (AZD9291) pemetrexed cisplatin or carboplatin
- Treatment Arm B (Placebo Comparator): All randomized patients will receive placebo QD with pemetrexed (500 mg/m^2) (with pre-treatment) plus either cisplatin (75 mg/m^2) or carboplatin (AUC5), both administered on Day 1 of 21-day cycles for 4 cycles, followed by placebo QD plus pemetrexed maintenance (500 mg/m^2) on Day 1 of 21-day cycles
  Interventions: Drug: Placebo for osimertinib (AZD9291) pemetrexed cisplatin or carboplatin

INTERVENTIONS:
Drug: Osimertinib (AZD9291) pemetrexed cisplatin or carboplatin — Randomized patients will receive oral dose of osimertinib with intravenous (IV) pemetrexed plus either IV cisplatin or IV carboplatin
  Arms: Treatment Arm A
Drug: Placebo for osimertinib (AZD9291) pemetrexed cisplatin or carboplatin — Randomized patients will receive oral dose of placebo matching osimertinib with IV pemetrexed plus either IV cisplatin or IV carboplatin
  Arms: Treatment Arm B

SUMMARY:
The study will evaluate the efficacy and safety of treatment with chemotherapy in combination with osimertinib compared to chemotherapy in combination with placebo in patients whose disease has progressed extracranially following first-line osimertinib treatment.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled study of platinum plus pemetrexed chemotherapy plus osimertinib versus platinum plus pemetrexed chemotherapy plus placebo in patients with epidermal growth factor receptor mutation-positive (EGFRm), locally advanced or metastatic NSCLC with or wihout stable brain metastases who responded to first-line osimertinib therapy (complete response [CR] or partial response [PR]) or stable disease (SD) for ≥ 6 months during first-line osimertinib treatment, and subsequently experienced radiological, extracranial disease progression. Approximately 204 patients were to be randomized in a 1:1 ratio to treatment with platinum plus pemetrexed chemotherapy plus osimertinib (Treatment Arm A) or platinum plus pemetrexed chemotherapy plus placebo (Treatment Arm B). However, the number of patients has been reduced to approximately 80 patients due to treatment landscape changes which outpaced study recruitment. Patients will be stratified based on the presence of brain metastases (stable brain metastases based on central nervous system (CNS) Response Evaluation Criteria in Solid Tumors, Version 1.1 [RECIST 1.1] assessments versus no brain metastases).

The 2 randomized treatment regimens are as follows:

* Treatment Arm A: Osimertinib 80 mg once daily (QD) with pemetrexed (500 mg/m^2) (with pre-treatment) plus either cisplatin (75 mg/m^2) or carboplatin (area under the concentration-time curve [AUC] 5), both administered on Day 1 of 21-day cycles for 4 cycles, followed by osimertinib 80 mg QD plus pemetrexed maintenance (500 mg/m^2) on Day 1 of 21-day cycles
* Treatment Arm B: Placebo QD with pemetrexed (500 mg/m^2) (with pre-treatment) plus either cisplatin (75 mg/m^2) or carboplatin (AUC5), both administered on Day 1 of 21-day cycles for 4 cycles, followed by placebo QD plus pemetrexed maintenance (500 mg/m^2) on Day 1 of 21-day cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
2. Pathologically confirmed non-squamous NSCLC.
3. Locally advanced (clinical stage IIIB or IIIC) or metastatic NSCLC (clinical stage IVA or IVB) or recurrent NSCLC, not amenable to curative surgery or radiotherapy.
4. Evidence of radiological extracranial disease progression following (Investigator-assessed) response or SD for ≥ 6 months during first-line osimertinib treatment, but who have not received further, subsequent treatment.
5. Tumor known to harbor 1 of the 2 or both common epidermal growth factor receptor (EGFR) mutations known to be associated with EGFR tyrosine kinase inhibitor (TKI) sensitivity (Ex19del or L858R), either alone or in combination with other EGFR mutations, which may include T790M.
6. World Health Organization performance status of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks.
7. Life expectancy >12 weeks at Day 1.
8. At least 1 lesion, not previously irradiated, that can be accurately measured.
9. Females must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of childbearing potential, or must have evidence of non-childbearing potential by fulfilling criteria at screening.
10. Male patients must be willing to use barrier contraception

Exclusion Criteria:

1. Clinical or radiological evidence of CNS progression on first-line osimertinib.
2. Past medical history of interstitial lung disease (ILD)/pneumonitis, drug-induced ILD/pneumonitis, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD/pneumonitis.
3. Any evidence of severe or uncontrolled systemic diseases.
4. Any of the following cardiac criteria:

   i) Mean resting QTc >470 msec ii) Any clinically important abnormalities in rhythm, conduction, or morphology of resting electrocardiogram iii) Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
5. Any concurrent and/or other active malignancy that has required treatment within 2 years of first dose of investigational product (IP).
6. Any unresolved toxicities from prior therapy.
7. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
8. More than 4 weeks elapsed since last dose of osimertinib by date of randomization.
9. Unable to tolerate osimertinib 80 mg first-line therapy.
10. Prior treatment with any systemic anti-cancer therapy.
11. Major surgery within 4 weeks of the first dose of IP.
12. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of IP.
13. Current use of medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP) 3A4.
14. Participation in another clinical study with an IP other than first-line osimertinib during the 4 weeks prior to Day 1.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-09-12 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2026-06-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (2):
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
- China (7):
  - Research Site, Beijing
  - Research Site, Ganzhou
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Zhengzhou
- Germany (4):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Hanover
  - Research Site, München
- Israel (5):
  - Research Site, Beersheba
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (8):
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Messina
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Terni
  - Research Site, Verona
- Spain (11):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Seville
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5162C00042&attachmentIdentifier=18187e36-5546-40ed-810d-6125a0239ad6&fileName=D5162C00042_PXL247131_Final_Draft_CSP__PDFA_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5162C00042&attachmentIdentifier=19604d92-3d31-425d-8aab-0a1a81e90c5b&fileName=D5162C00042_PXL247131_Final_Draft__SAP_PDFA_redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5162C00042&attachmentIdentifier=baec234a-e181-4ed0-9ce5-2a9e6798c476&fileName=D5162C00042_PXL247131_Final_Draft_CSR_synopsis_PDFA_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 12 September 2021 (First participant in) and the analyses presented in this results form are based on a final data cut-off of 28 October 2024.
Pre-assignment Details: Participants meeting eligibility criteria predefined in protocol were enrolled in the study. Assessments performed as per the schedule of the assessments.
Groups:
- Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin: Participants received osimertinib 80 mg once daily (QD) with pemetrexed (500 mg/m2) (with pre-treatment) plus either cisplatin (75 mg/m2) or carboplatin, both administered on Day 1 of 21-day cycles for 4 cycles, followed by osimertinib 80 mg QD plus pemetrexed maintenance (500 mg/m2) on Day 1 of 21-day cycles.
- Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin: Participants received placebo QD with pemetrexed (500 mg/m2) (with pre-treatment) plus either cisplatin (75 mg/m2) or carboplatin, both administered on Day 1 of 21-day cycles for 4 cycles, followed by placebo QD plus pemetrexed maintenance (500 mg/m2) on Day 1 of 21-day cycles.
Period: Overall Study
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin
Started | 49 | 49
Completed | 0 | 0
Not Completed | 49 | 49
Not completed — Failure to meet randomization criteria | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 25 | 28
Not completed — Participants ongoing study at data cutoff date of 28-Oct-24 | 21 | 16

BASELINE CHARACTERISTICS:
Population: The full analysis set consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (11.39) | 61.0 (10.02) | 61.5 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 39 | 69
  Male | 19 | 10 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 45 | 42 | 87
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as time from randomization until progression (intracranial or extracranial, whichever occurs first) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (for extracranial progression) and Central nervous system (CNS) RECIST 1.1 (for intracranial progression) as assessed by the Investigator at local site or death due to any cause.
Time Frame: From date of first dose (Day 1) until date of progression at local site or death due to any cause or data cut-off date whichever occurred first (up to 3 years 1 month)
Population: The Full analysis set consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin
Number analyzed (Participants) | 49 | 49
Months | 8.4 [5.75 to 11.83] | 4.4 [3.52 to 5.55]

2. Secondary Outcome: Intracranial Progression Free Survival With Brain Metastases at Baseline
Description: Intracranial PFS (IC-PFS) is defined as time from randomization until intracranial progression per CNS RECIST 1.1 as assessed by the Investigator at local site or death due to any cause.
  For participants with brain metastases at baseline, the IC-PFS rate at specified timepoints was estimated using the Kaplan-Meier method which indicated the percentage of these participants who remain alive and free from intracranial progression per CNS RECIST 1.1 as assessed by the Investigator. The data was calculated throughout the study as per the below timeframe but IC-PFS rate at 6 months has been presented as it was clinically relevant.
Time Frame: Assessed from date of first dose (Day 1) until date of intracranial progression at local site or death due to any cause or data cut off date whichever occurred first (up to 3 years 1 month), data for 6 months reported
Population: The Full analysis set consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin
Number analyzed (Participants) | 11 | 12
Percentage of participants | 81.8 [44.74 to 95.12] | 55.6 [20.42 to 80.45]

3. Secondary Outcome: Intracranial Progression Free Survival Without Brain Metastases at Baseline
Description: Intracranial PFS (IC-PFS) is defined as time from randomization until intracranial progression per CNS RECIST 1.1 as assessed by the Investigator at local site or death due to any cause.
  For participants without brain metastases at baseline, the IC-PFS rate at specified timepoints was estimated using the Kaplan-Meier method which indicated the percentage of these participants who remain alive and free from intracranial progression per CNS RECIST 1.1 as assessed by the Investigator. The data was calculated throughout the study as per the below timeframe but IC-PFS rate at 6 months has been presented as it was clinically relevant.
Time Frame: as for outcome 2
Population: The Full analysis set consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin
Number analyzed (Participants) | 38 | 37
Percentage of participants | 86.7 [68.08 to 94.83] | 63.1 [42.87 to 77.81]

4. Secondary Outcome: Extracranial Progression Free-survival
Description: Extracranial PFS is defined as time from randomization until extracranial progression per RECIST 1.1 as assessed by the Investigator at local site or death due to any cause.
Time Frame: From date of first dose (Day 1) until date of extracranial progression at local site or death due to any cause or data cut-off date whichever occurred first (up to 3 years 1 month)
Population: The Full analysis set consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin
Number analyzed (Participants) | 49 | 49
Months | 8.4 [5.75 to 11.83] | 5.2 [3.52 to 5.78]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the length of time from randomization until the date of death due to any cause.
Time Frame: From date of first dose (Day 1) until post progression survival follow-up (up to 3 years 1 month)
Population: The Full analysis set consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin
Number analyzed (Participants) | 49 | 49
Months | 15.9 [12.39 to 20.83] | 9.8 [8.38 to 17.25]

ADVERSE EVENTS:
Time Frame: From date of first dose (Day 1) until Follow-up (28 days post last dose) (up to 3 years 1 month)
Description: The safety analysis set consisted of all randomized participants who had received at least 1 dose of IP.
Arm/Group | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin
All-Cause Mortality (participants affected / at risk) | 26/48 | 28/48
Serious Adverse Events (participants affected / at risk) | 18/48 | 15/48
Other Adverse Events (participants affected / at risk) | 46/48 | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin (N=48) | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin (N=48)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Right hemisphere deficit syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm A: Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin (N=48) | Treatment Arm B: Placebo for Osimertinib (AZD9291), Pemetrexed, Cisplatin or Carboplatin (N=48)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 7 (7) | 2 (2)
COVID-19 (Infections and infestations) | 6 (6) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Paronychia (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 30 (64) | 26 (44)
Leukocytosis (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (7) | 4 (8)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 10 (22) | 9 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (11) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 8 (16) | 9 (11)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypoalbuminaemi (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (8)
Dysgeusia (Nervous system disorders) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 3 (3)
Paraesthesia (Nervous system disorders) | 4 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (6) | 4 (6)
Constipation (Gastrointestinal disorders) | 11 (12) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 15 (19) | 5 (6)
Nausea (Gastrointestinal disorders) | 17 (37) | 23 (43)
Stomatitis (Gastrointestinal disorders) | 5 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 13 (18) | 9 (24)
Hepatotoxicity (Hepatobiliary disorders) | 3 (3) | 1 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 (6) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 19 (40) | 23 (40)
Fatigue (General disorders) | 5 (12) | 3 (4)
Oedema peripheral (General disorders) | 6 (8) | 4 (7)
Pyrexia (General disorders) | 6 (7) | 3 (3)
Alanine aminotransferase increased (Investigations) | 8 (13) | 9 (15)
Aspartate aminotransferase increased (Investigations) | 7 (10) | 7 (14)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 5 (6)
Blood creatinine increased (Investigations) | 8 (13) | 4 (7)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (4) | 5 (7)
Lymphocyte count decreased (Investigations) | 2 (4) | 4 (8)
Neutrophil count decreased (Investigations) | 9 (39) | 12 (22)
Platelet count decreased (Investigations) | 10 (21) | 2 (3)
White blood cell count decreased (Investigations) | 6 (31) | 8 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (2):
  • Study Protocol (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT04765059/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04765059/SAP_001.pdf